CLINICAL TRIAL: NCT05851365
Title: A Pilot Study of Magnetic Resonance (MR) Imaging With Hyperpolarized Bicarbonate (13C) to Measure Tissue pH in Localized Prostate Cancer
Brief Title: Magnetic Resonance (MR) Imaging With Hyperpolarized Bicarbonate (13C) to Measure Tissue pH in Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Robert Flavell, MD, PhD (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Robert Flavell, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23922; NCI-2023-03218 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Localized Prostate Carcinoma
Keywords: Tissue pH; Magnetic Resonance (MR) Imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-surgical participants with prostate cancer (Experimental): The hyperpolarized 13C bicarbonate injection includes the administration of 35 mL injected intravenously (IV) at a rate of 5 mL/second followed by a 20 mL saline flush at 5 mL/second, followed by magnetic resonance (MR) imaging. The intervention will include routine and safety assessments 5 to 9 days after the injection.
  Interventions: Drug: Hyperpolarized Bicarbonate (13C); Procedure: Magnetic Resonance imaging

INTERVENTIONS:
Drug: Hyperpolarized Bicarbonate (13C) — Given IV
  Other Names: Hyperpolarized (HP) bicarbonate 13 (13C); HP C13
Procedure: Magnetic Resonance imaging — Magnetic resonance imaging is a medical imaging technique used in radiology to form pictures of the anatomy and the physiological processes of the body
  Other Names: Magnetic Resonance scan; MR scan

SUMMARY:
This is a single site, prospective pilot study to determine the feasibility and safety of the administration of HP 13C bicarbonate in 10 patients with prostate cancer to determine potential hydrogen (pH) values in surrounding tissue. The proposed study will evaluate pre-surgical participants with histologically confirmed localized prostate cancer who receive infusion of hyperpolarized 13C injection prior to MR imaging with endorectal coil.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of tumor pH measurement in men with prostate cancer using hyperpolarized 13C bicarbonate imaging.

SECONDARY OBJECTIVE:

I. To determine the safety of administration of hyperpolarized 13C-bicarbonate.

EXPLORATORY OBJECTIVES:

I. To correlate the measurement of tissue pH with pathologic grade.

II. To correlate tissue pH maps with immunohistochemistry staining (IHC), gene expression (RNA-Seq), and spatial transcriptomics. *Bristol Myers Squibb (BMS) collaboration

OUTLINE:

Men with biopsy-proven adenocarcinoma of the prostate scheduled to undergo radical prostatectomy at University of California, San Francisco (UCSF) within 12 weeks of enrollment will receive infusion with hyperpolarized 13C bicarbonate and undergo metabolic MR imaging with endorectal coil. Participants will be followed for 5-9 days after the hyperpolarized 13C-bicarbonate injection, or removal from study, or until death, whichever occurs first. Participants removed from study for unacceptable study related adverse event(s) will be followed until resolution or stabilization (as determined by the investigator) or until initiation of new anti-cancer therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age >=18 years.
2. Patients must have biopsy-proven adenocarcinoma of the prostate; biopsy may be performed outside of University of California, San Francisco (UCSF) if detailed results of sextant biopsy are available.
3. Tumor size of at least 1.0 cm in long axis on Magnetic resonance imaging (MRI) or ultrasound; if no prior imaging is available, at least 3 cores positive on biopsy.
4. Patients must have planned radical prostatectomy at UCSF within 12 weeks following protocol MRI/ magnetic resonance spectroscopy imaging) (MRSI).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Demonstrates adequate organ function as defined below:

   1. Adequate bone marrow function:

      * Absolute neutrophil count >=1,500 cells/µL.
      * Platelets >=75,000 cells/µL.
      * Hemoglobin >=9.0 gm/dL.
   2. Adequate hepatic function:

      * Total bilirubin <1.5x upper limits of normal (ULN) (within normal institutional limits, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits).
      * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) <=1.5 X institutional upper limit of normal.
      * Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <=1.5 X institutional upper limit of normal.
   3. Adequate renal function:

      * Creatinine clearance >= 50 calculated using the Cockcroft-Gault equation, unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who because of general medical or psychiatric condition, or physiologic status, cannot give valid informed consent.
2. Patients unwilling or unable to undergo MR imaging, including patients with contraindications to Magnetic resonance imaging (MRI) as per UCSF radiology departmental guidelines.
3. Patients who cannot tolerate or have contra-indications to endorectal coil insertion, for example, patients with a prior abdominoperineal resection of the rectum or latex allergy.
4. Patients with contra-indications to injection of gadolinium contrast as per UCSF radiology departmental guidelines.
5. Patients who take carbonic anhydrase inhibitors (e.g. acetazolamide, dichlorphenamide, methazolamide).
6. Metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging.
7. Cryosurgery, surgery for prostate cancer, prostatic or pelvic radiotherapy prior to study enrollment. No limit on number of prior prostate biopsies. Prior Transurethral Resection of the Prostate (TURP) is not allowed.
8. Poorly controlled hypertension, with blood pressure at study entry >160/100. The addition of anti-hypertensives to control blood pressure is allowed for eligibility determination.
9. Congestive heart failure or New York Heart Association (NYHA) status >= 2. A history of clinically significant electrocardiogram (EKG) abnormalities, including QT prolongation, a family history of prolonged QT interval syndrome, or myocardial infarction (MI) within 6 months of study entry. Patients with rate-controlled atrial fibrillation/flutter will be allowed on study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a signal to noise ratio > 2 | Day of MR imaging (1 day)
  The feasibility of a study will be determined by the ability to generate adequate signal to noise ratio to measure acidity (pH) in tumor or adjacent healthy tissue. This study will be considered successful if the 13C bicarbonate (CO2) and 13C-CO2 resonances in tumor or normal prostate are qualitatively detectable and signal to noise ratios are greater than 2. The point estimation and 95% confidence intervals (CI) of the participants having sufficient signal to noise ratio will be obtained using the Wilson Score confidence interval method.

SECONDARY OUTCOMES:
Percentage of participants with reported treatment-emergent adverse events | Up to 9 days
  To assess the safety of the administration of hyperpolarized 13C bicarbonate; adverse events will be collected and recorded by type, severity (grade) and attribution according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The percentage of participants with grade 2 and higher, treatment-emergent adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Flavell, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No